CLINICAL TRIAL: NCT04195763
Title: A Prospective Study to Evaluate the Patient Reported Quality of Life Prior to and After Strensiq® Treatment in Adults With Pediatric Onset Hypophosphatasia
Brief Title: Patient Reported Outcomes in Adults With Pediatric-onset Hypophosphatasia Treated With Strensiq® (Asfotase Alfa)
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Xcenda, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: ALX-HPP-503
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Hypophosphatasia
Keywords: Pediatric-onset hypophosphatasia; Pediatric-onset; Hypophosphatasia; HPP; Patient reported outcome
MeSH Terms: conditions — Hypophosphatasia | interventions — asfotase alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Pediatric-onset HPP: Adult participants diagnosed with pediatric-onset HPP, newly prescribed treatment with asfotase alfa, and registered in the patient support program managed by OneSource.
  Interventions: Drug: asfotase alfa

INTERVENTIONS:
Drug: asfotase alfa — This is an observational study and no intervention will be administered. All participants will be treated by their physician in accordance with standard of care. All medications are commercially available and will be used as directed by the treating physician.
  Other Names: Strensiq®

SUMMARY:
This observational study will evaluate the treatment effect of Strensiq (asfotase alfa) on Patient Reported Outcomes (PROs) in participants diagnosed with pediatric-onset hypophosphatasia (HPP) registered in the patient support program managed by OneSource™.

DETAILED DESCRIPTION:
Participants consenting to participate in this study will be asked to complete study questionnaires by phone interviews upon consenting (Baseline), and up to 12 months following treatment initiation with asfotase alfa. Demographic and clinical characteristics of participants in the study will be characterized.

This is an observational study and no intervention will be administered. Participants will be treated in accordance with standard of care.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Clinical diagnosis of pediatric-onset HPP
* Naïve to asfotase alfa
* Expected to begin treatment with asfotase alfa for HPP
* Registered in OneSource
* Willing and able to provide voluntary, verbal informed consent to participate in this study

Exclusion Criteria:

* Pregnant or breastfeeding
* Unable to speak and understand English
* Unable or unwilling to complete the study surveys via telephone interview at the protocol-required time points

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female participants ≥18 years of age who have been diagnosed with pediatric-onset HPP, have been newly prescribed treatment with asfotase alfa, and are registered in the patient support program managed by OneSource will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline In Patient Reported Outcomes (PROs) Questionnaire Scores | Baseline, up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xcenda, LLC, Palm Harbor, Florida, United States

IPD SHARING:
Plan to Share IPD: No